CLINICAL TRIAL: NCT02590783
Title: Treatment of Pelvic Ring Fractures in the Elderly: A Randomized Controlled Trial Comparing Surgical vs. Conservative Therapy
Brief Title: Treatment of Pelvic Ring Fractures in the Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study question was not suitable
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-188
Record Dates: First submitted 2015-09-22; First posted 2015-10-29 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Pain
Keywords: treatment
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental intervention surgery (Experimental): screw osteosynthesis of the sacrum and in certain cases additional plate osteosynthesis of dislocated pubic rami fractures, postoperative analgesia, physiotherapy, work-up for osteoporosis, geriatric rehabilitation if necessary
  Interventions: Procedure: experimental intervention surgery
- control intervention conservative (Active Comparator): analgesia, physiotherapy, work-up for osteoporosis, geriatric rehabilitation if necessary
  Interventions: Procedure: control intervention

INTERVENTIONS:
Procedure: experimental intervention surgery — Patients are placed supine on the carbon table. Screw paths are planned on a spiral CT scan from the sacrum on transversal slices, two Kirschner-wires 2.5 mm in diameter are introduced into the iliac bone through a stab incision and advanced into the ilio-sacral joint, through the lateral part of sacrum into the first and second sacral body, through the contralateral lateral part of the sacrum and exiting the contralateral iliac bone through the sacra-iliac joint with aid of CT-guidance. Over the Kirschner-wires 7.0 mm cannulated screws are introduced and the Kirschner-wires withdrawn. Several low-dose computer tomography scans are performed to secure the correct position. Total radiation dose is 300 mille gray square centimetres (mGycm).
  Arms: experimental intervention surgery
Procedure: control intervention — Mobilization guided by our physiotherapists. Full weight bearing is allowed. Analgetic treatment with metamizol, ibuprofen or paracetamol to the attending physicians discretion under regular surveillance laboratory values and/ or morphine or methadone. Patients will be treated with an individually based approach, if necessary involving our anesthesiologic pain service. Thrombo-embolic prophylaxis with a low molecular weight heparin or rivaroxaban for 6 weeks unless there is an indication for oral anticoagulation. All patients will be followed up by the Geriatric Fracture Center considering osteoporosis, fall prophylaxis, malnutrition and delirium. For the duration of the study the patients will not receive Parathyroid Hormone Substitution or Phosphonates.
  Arms: control intervention conservative

SUMMARY:
Pelvic ring fractures in the elderly are associated with high morbidity during standard conservative treatment due to immobility. Furthermore the risk of long term dependence even after the fracture has united is high. In analogy to the treatment of hip fractures in a similar patient population, patients might benefit from surgical treatment due to a reduction in pain and early mobilization.

DETAILED DESCRIPTION:
Comparison of surgical vs conservative treatment with respect to mobility, pain, morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* CTI/MRI verified fracture of the sacrum affecting the posterior ring or both posterior and anterior ring
* age>65 years, ambulatory with/without walking aids before Trauma
* ambulatory with/without walking aids before trauma
* postmenopausal status in women
* informed consent for study participation and surgery

Exclusion Criteria:

* Refusal of consent by the patient or legal representatives to participate in the study
* Other fractures or
* Unstable pelvic fracture (type B or C according to classification of 'Arbeitsgemeinschaft für Osteosynthesefragen' (AO)/OTA) requiring surgical stabilisation after high- or low-energy trauma
* Suspicion of a pathological fracture in the context of known or unknown malignancy
* Previous surgery of the pelvis with metal obstructing the planned paths of the ilio-sacral screws
* Symptomatic low back pain with morphological changes, i.e. intervertebral disc displacement, neoplasm metastasis in the axial skeleton, spinal stenosis, vertebral fracture, spondylarthropathy etc.
* Comorbidity that precludes undergoing general or spinal anaesthesia
* Pre-trauma mobility status that precludes achieving a post-trauma mobility status enabling the patient to perform the timed up and go test (e.g. patient being in a wheel chair)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Mobility at 3 weeks post-diagnosis | 3 weeks post-diagnosis
  Quality of mobilization will be compared using the TUG test. The primary endpoint is TUG at 3 weeks following diagnosis (+/- 3 days) all TUG measurements are assessed by the study nurse.

SECONDARY OUTCOMES:
Activities of Daily Living (ADL) at baseline | baseline
  Functional recovery will be measured using the ADL score.
Activities of Daily Living (ADL) at 4-7 days after diagnosis | 4-7 days after diagnosis
  Functional recovery will be measured using the ADL score.
Activities of Daily Living (ADL) at 3 weeks | 3 weeks
  Functional recovery will be measured using the ADL score.
Activities of Daily Living (ADL) at 3 months | 3 months
  Functional recovery will be measured using the ADL score.
Activities of Daily Living (ADL) at 12 months | 12 months
  Functional recovery will be measured using the ADL score.
Pain (VAS 10) at baseline | baseline
  Pain will be assessed using the 10 point Visual Analogue Scale (VAS10).
Pain (VAS 10) at 4-7 days after diagnosis | 4-7 days after diagnosis
  Pain will be assessed using the 10 point Visual Analogue Scale (VAS10).
Pain (VAS 10) at 3 weeks | 3 weeks
  Pain will be assessed using the 10 point Visual Analogue Scale (VAS10).
Pain (VAS 10) at 3 months | 3 months
  Pain will be assessed using the 10 point Visual Analogue Scale (VAS10).
Number of patients that are able to return to their pre-injury living situation at 3 months | 3 months
  Number of patients that are able to return to their pre-injury living Situation. The outcome to compare the "return to the pre-injury living situation".
Number of patients that are able to return to their pre-injury living situation at 12 months | 12 months
  Number of patients that are able to return to their pre-injury living Situation. The outcome to compare the "return to the pre-injury living situation".

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Jakob, Prof, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Rommens PM, Hofmann A. Comprehensive classification of fragility fractures of the pelvic ring: Recommendations for surgical treatment. Injury. 2013 Dec;44(12):1733-44. doi: 10.1016/j.injury.2013.06.023. Epub 2013 Jul 18. PMID 23871193